CLINICAL TRIAL: NCT03844373
Title: Tolerance and Acceptability Evaluation of STOCKHOLM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AY:APL:OPD
Record Dates: First submitted 2019-02-06; First posted 2019-02-18 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — antithrombin III Stockholm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients established on an oral nutritional supplement, being prescribed oral nutritional supplement (ONS) providing at least 300 kcal/day will be changed onto an equivalent prescription of STOCKHOLM for a period of 9 days.
  Interventions: Dietary Supplement: STOCKHOLM

INTERVENTIONS:
Dietary Supplement: STOCKHOLM — STOCKHOLM is a Food for Special Medical Purposes (FSMP) and must, therefore, be used under medical supervision.

SUMMARY:
Tolerance and Acceptability of new oral nutritional supplement - STOCKHOLM.

DETAILED DESCRIPTION:
To evaluate tolerance and acceptability of 'STOCKHOLM' in patients requiring supplementary oral nutritional support compared with currently available alternatives.

To obtain data to support an ACBS submissions for 'STOCKHOLM' (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to communicate their views regarding acceptability.
* Patients established on an oral nutritional supplement, being prescribed ONS providing approximately 300 kcal/day
* Patients expected to require oral nutritional supplementation for at least 2 further weeks.
* Informed consent obtained.

Exclusion Criteria:

* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Patients requiring a milk free diet
* Patients with medical or dietary contraindication to any feed ingredients (see appendix 2 of protocol for full list)
* Patients with significant renal or hepatic impairment
* Patients with dysphagia requiring stage 1,2 or 3 thickened fluids
* Patients with uncontrolled inflammatory bowel disease or previous bowel resection with ongoing gastrointestinal symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
GI Tolerance | 9 Days
  To assess gastro-intestinal tolerance of 'STOCKHOLM' in patients in the community requiring oral nutritional supplementation. Monitoring includes recording the number and consistency of bowel movements as assessed on the Bristol stool form scale, any episodes of nausea, vomiting, abdominal pain, bloating or diarrhoea.

SECONDARY OUTCOMES:
Acceptability and Palatability of Consuming the Nutritional Supplement: Questionnaire | 9 days
  To assess the acceptability of 'STOCKHOLM' in patients in the community requiring oral nutritional supplementation. At the end of the intervention period an acceptability and preference questionnaire will be completed by the patient in order to seek their opinion on the taste, smell, texture and overall liking of the new supplement drink.
Compliance with Prescription of STOCKHOLM | 9 days
  Recording of amount of STOCKHOLM consumed by subjects compared to amount prescribed. Good compliance = >80% of prescribed being consumed. Same data collected for baseline product and compared with that of STOCKHOLM.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma Fry, Haywards Heath, United Kingdom

IPD SHARING:
Plan to Share IPD: No